CLINICAL TRIAL: NCT02282787
Title: DEXMEDETOMIDINE ADJUVANT TO LOCAL ANAESTHESIA FOR PERIBULBAR BLOCKS IN RETINAL SURGERY
Brief Title: Dexmedetomidine Adjuvant in Retinal Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Marwan Abouammoh, Associate professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: E-14-1291
Record Dates: First submitted 2014-10-31; First posted 2014-11-04 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Peribulbar Anesthesia
Keywords: local anesthesia; peribulbar anesthesia; DEXMEDETOMIDINE; vitreoretinal surgery
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5 micron dex arm (Experimental)
  Interventions: Drug: DEXMEDETOMIDINE
- 10 micron dex arm (Experimental)
  Interventions: Drug: DEXMEDETOMIDINE

INTERVENTIONS:
Drug: DEXMEDETOMIDINE — Does adding 5 or 10 micron of DEXMEDETOMIDINE to peribulbar anesthesia is any different from regular peribulbar anesthesia practice?

SUMMARY:
During LA in retinal surgery there is some problem as regard the lack of anaesthesia duration and unexpected globe movement .so many adjuvant was added to LA to overcome this disadvantages of LA such as clonidine and fentanyl .

The investigators hypothesis is adding dexmedetomidine to pribulbal blocking LA will prolong anaesthesia duration and improve globe akinesia and decrease intraoperative supplementation of LA.There are Many studies had described the effects of dexmedetomidine on peripheral nerve blocks, spinal but up to date no knowledge is available on the impact of dexmedetomidine adjuvant to local anaesthetic in ophthalmic surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Going for elective vitreoretinal surgery.

Exclusion Criteria:

* History of coagulation abnormalities.
* Allergy to local anesthetics.
* Cardiac, hepatic or renal failure,
* Chronic clonidine or analgesic therapy.
* One-eyed patients

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
onset, duration of the motor and sensory block | 10 minutes from injection
  A block was considered satisfactory when complete akinesia occurred. In the absence of complete akinesia in any direction after 10 min, supplementary anesthesia given by a further injection of 2-4 ml of the test solution in the same manner as given before. Calculate the number of patients needed supplemental block were. The surgeon assessed the duration of surgery anesthesia and akinesia. Intraocular pressure measured before block, immediately after block and before surgical procedures

SECONDARY OUTCOMES:
observe the adverse effects of Dexmedetomidine | during and after surgery
  ECG, invasive BP and pulse oximetry will apply to all patients.
  • The haemodynamic parameters (MAP and HR) will be continuously measured, and will be recorded at before induction (baseline), one minute after block . after 5 minutes then at the surgical incision, 15-min intervals intraoperatively, the end of surgery and10 and 20 minutes postoperatively.
  Incidence of Oculocardiac reflex (OCR) or any arrhythmia during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Abouammoh, MD, Principal Investigator — King Saud University
Locations (1):
- King Abdulaziz University Hospital at King Saud University, Riyadh, Riyadh Region, Saudi Arabia